CLINICAL TRIAL: NCT01801371
Title: Diagnostic Performance and Evaluation Efficacy of Brain 68Ga-BNOTA-PRGD2 PET/CT in Pre-surgery Glioma Patients
Brief Title: 68Ga-BNOTA-PRGD2 PET/CT in Diagnosis and Evaluation of Glioma
Acronym: GRGDG
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhaohui Zhu, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM6
Record Dates: First submitted 2013-02-22; First posted 2013-02-28 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Glioma
Keywords: Glioma; Diagnostic imaging; Integrin receptor; 68Ga-BNOTA-PRGD2; PET/CT
MeSH Terms: conditions — Glioma | interventions — 68gallium-BNOTA-PRGD2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-BNOTA-PRGD2 (Experimental): In patients in suspicion of glioma, single bolus of nearly 111 MBq 68Ga-BNOTA-PRGD2 will be intravenously injected 30 minutes before brain PET/CT to determine 68Ga-BNOTA-PRGD2 uptake in tumor and brain.
  Interventions: Drug: 68Ga-BNOTA-PRGD2

INTERVENTIONS:
Drug: 68Ga-BNOTA-PRGD2 — Single intravenous bolus injection of nearly 111 MBq 68Ga-BNOTA-PRGD2 at 30 minutes before brain PET/CT scanning.
  Other Names: 68Ga-p-SCN-Bn-NOTA-PEG3-RGD2

SUMMARY:
This is an open-label brain PET/CT (positron emission tomography/computed tomography) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-BNOTA-PRGD2 in glioma patients. A single dose of nearly 111 MBq 68Ga-BNOTA-PRGD2 (≤40 µg BNOTA-PRGD2) will be intravenously injected into patients in suspicion of glioma. Visual and semiquantitative method will be used to assess the PET/CT images. Brain MRI with/without enhancement and 18F-FDG PET/CT will be performed for comparison. The postoperative pathology and integrin αvβ3 and CD34 immunohistochemical stains will also be used for correlation.

DETAILED DESCRIPTION:
Integrin αvβ3 is an important member of integrin receptor family and expressed preferentially on various types of tumor cells and the activated endothelial cells of tumor angiogenesis, but not or very low on the quiescent vessel cells and other normal cells. Therefore, the integrin αvβ3 receptor is becoming a valuable target for diagnosis and response evaluation of malignant tumors.

The tri-peptide sequence of arginine-glycine-aspartic acid (RGD) can specifically bind to the integrin αvβ3 receptor. Accordingly, a variety of radio-labeled RGD-based peptides have been developed for non-invasive imaging of integrin αvβ3 receptor expression via positron emission tomography (PET) or single photon emission computed tomography (SPECT). Among all RGD radiotracers, several PET imaging agents, including 18F-Galacto-RGD and 18F-AH111585, have been investigated in clinical trials for tumor diagnosis, and the results demonstrated that both radiotracers allowed the specific imaging of various types of tumors, and the tumor uptake correlated well with the expression of integrin αvβ3. Recently, serial RGD dimeric peptides with PEG linkers have been studied. The new types of RGD peptides showed much higher in vitro integrin αvβ3-binding affinity than the single RGD tri-peptide sequence, and importantly, they exhibited significantly increased tumor uptake and improved in vivo kinetics in animal models. As a representative, 68Ga-BNOTA-PRGD2 could be easily prepared and exhibited excellent in vivo behaviors in animal models. No adverse reactions have been observed in animal models to date.

For the further interests in clinical translation of 68Ga-BNOTA-PRGD2, an open-label brain PET/CT study was designed to investigate the diagnostic performance and evaluation efficacy of 68Ga-BNOTA-PRGD2 in pre-surgery glioma patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥18 years old；
* In suspicion of brain glioma on MRI；
* The tumor will be surgically removed and histological diagnosis will be available.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential；
* Known severe allergy or hypersensitivity to IV radiographic contrast；
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Semiquantitative measurement of standardized uptake values (SUVs) of lesions | 1 year
  The semiquantitative analysis will be performed by the same person for all cases, and the standardized uptake value (SUV) of each tumor will be measured using a volume of interest (VOI) method.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety | 1 year
  Adverse events within 5 days after 68Ga-BNOTA-PRGD2 injection and PET/CT scanning will be collected and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No